CLINICAL TRIAL: NCT05368272
Title: EEG Spectrogram to Assess Brain Vulnerability as a Risk Factor for Postoperative Delirium in Older People - a Feasibility Study
Brief Title: EEG Spectrogram, Brain Vulnerability and POD
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21074
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Delirium
Keywords: processed EEG; Postoperative vulnerability; Older people; Brain vulnerability
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Processed electroencephalography — Acquisition of raw EEG data from processed EEG monitor. Analysis of data acquired for prespecified bandwidth properties
Other: Postoperative delirium assessment — Twice daily assessment for the incidence of postoperative delirium using validated tool (questionnaire)

SUMMARY:
An assessment of difference in prespecified processed electroencephalography variables between cognitively intact older surgical patients who develop postoperative delirium compared to those who do not develop postoperative delirium

DETAILED DESCRIPTION:
Postoperative delirium in older people may be contributed to by intrinsic brain vulnerability such as pre-existing dementia. Some cognitively intact older people also experience postoperative delirium and in these patients some go on to develop later dementia. The investigators propose that postoperative delirium may be an unmasking of covert brain vulnerability by the dyshomeostasis of the anaesthesia/surgical intervention.

In people with dementia or mild cognitive impairment, electroencephalography (EEG) studies have shown slowing of brain wave activity, especially in the back of the brain.

Processed electroencephalography, using a limited number of channels, is routinely used during anaesthesia to aid assessment of anaesthetic depth of the patient.

In this study the investigators will assess the feasibility of acquiring EEG data from the front and back of the brain. The investigators will also explore the data for early signals of brain vulnerability

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Elective, moderate/major, non-neuro, non-cardiac surgery
* Ability to give informed consent

Exclusion Criteria:

* Preoperative cognitive impairment
* Current systemic infection
* Current use of medication that may modify EEG
* History of neurosurgery/significant head trauma
* Presence of neurological diseases including overt stroke, dementia, epilepsy, multiple sclerosis, Parkinson's disease, intracranial tumours and other significant neurologic disorders
* Current significant psychiatric conditions such as severe depression.
* Palliative surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older people scheduled for elective major surgery at a large teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of acquiring frontal and posterior EEG data from the Narcotrend monitor during the preoperative and intraoperative period | Approximately 1 - 2 hours per participant
  Feasibility will be assessed by the ability to get preoperative and intraoperative epochs of EEG that clearly demonstrates the different brain wave bands (alpha, theta and delta)

SECONDARY OUTCOMES:
Preoperative brain wave differences | Approximately 10 minutes per participant
  Identify any differences in frontal and posterior narrowband (i.e. alpha, delta and theta) power preoperatively between older people who develop POD compared to those who do not.
Change in brain wave power due to induction of anaesthesia | Approximately 1 hour per particpant
  Identify if the change in narrowband power from the preoperative values to steady state intraoperative values are different between groups (i.e. people who develop POD vs people who do not develop POD)
Intraoperative brain wave patterns | Duration of surgery or 2 hours (shortest option)
  Identify any differences in mean and spectral edge frequencies preoperatively and intraoperatively between older people who develop POD and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Iain Moppett, FRCA, MD, Principal Investigator — University of Nottingham
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No